CLINICAL TRIAL: NCT04162769
Title: A Multicenter, Randomized, Double-Blinded, Placebo-Controlled 16-Week Study (With a 52-Week Open-Label Extension) to Assess the Safety and Efficacy of Etrasimod in Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study to Assess the Safety and Efficacy of Etrasimod in Subjects With Moderate-to-Severe Atopic Dermatitis
Acronym: ADVISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APD334-201
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Atopic Dermatitis
Keywords: Moderate-to-severe atopic dermatitis; Etrasimod; APD334
MeSH Terms: conditions — Dermatitis, Atopic | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 12-Week Double-Blind Treatment Period: Etrasimod 1 milligrams (mg) (Experimental)
  Interventions: Drug: Etrasimod 1 mg
- 12-Week Double-Blind Treatment Period: Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod 2 mg
- 12-Week Double-Blind Treatment Period: Placebo (Placebo Comparator)
  Interventions: Drug: Etrasimod matching placebo
- 52-Week Open-Label Extension Period: Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod 2 mg

INTERVENTIONS:
Drug: Etrasimod 1 mg — Etrasimod 1 mg tablet taken by mouth, once daily
  Other Names: APD334
  Arms: 12-Week Double-Blind Treatment Period: Etrasimod 1 milligrams (mg)
Drug: Etrasimod 2 mg — Etrasimod 2 mg tablet taken by mouth, once daily.
  Other Names: APD334
  Arms: 12-Week Double-Blind Treatment Period: Etrasimod 2 mg; 52-Week Open-Label Extension Period: Etrasimod 2 mg
Drug: Etrasimod matching placebo — Etrasimod matching placebo tablet by mouth, once daily.
  Arms: 12-Week Double-Blind Treatment Period: Placebo

SUMMARY:
The purpose of this study is to determine whether etrasimod is a safe and effective treatment for moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion criteria:

* Participants with chronic atopic dermatitis, defined by Hanifin and Rajka criteria, that has been present for at least 1 year prior to the Screening Visit
* Participants with Eczema Area and Severity Index (EASI) ≥ 12 at the Screening Visit and ≥ 16 at the Baseline Visit
* Participants with validated Investigator's Global Assessment (vIGA) score ≥ 3 (on the 0 to 4 vIGA scale, in which 3 = moderate and 4 = severe) involvement at the Screening and Baseline visits

Exclusion Criteria:

* Presence of skin comorbidities that would interfere with study assessments of the underlying disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (38):
- United States (35):
  - Noble Clinical Research, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - First OC Dermatology, Fountain Valley, California
  - Marvel Research LLC, Huntington Beach, California
  - ADVA Clinical Research, Inc, Inglewood, California
  - Providence Clinical Research, North Hollywood, California
  - TCR Medical Corporation, San Diego, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Prohealth Research Center, Doral, Florida
  - Aby's New Generation Research, Inc., Hialeah, Florida
  - Skin Care Research, LLC, Hollywood, Florida
  - Advanced Research Institute of Miami LLC, Homestead, Florida
  - Amber Pediatrics Research, LLC, Homestead, Florida
  - South Miami Medical & Research Group. Inc, Miami, Florida
  - Amber Pediatrics Research, LLC, Miami, Florida
  - Skin Research of South Florida, Miami, Florida
  - Amber Clinical Research, LLC, Miami Shores, Florida
  - IMA Clinical Research, LLC, St. Petersburg, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Skin Sciences PLLC, Louisville, Kentucky
  - Quinn Healthcare/SKYCRNG, Ridgeland, Mississippi
  - Quality Clinical Research Inc, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Greenwich Village Dermatology, New York, New York
  - ODRC Enterprises, LLC dba Oregon Dermatology and Research Center, Portland, Oregon
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Gadolin Research, Beaumont, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - FMC Science, Georgetown, Texas
  - FMC Science, Lampasas, Texas
  - Alliance for Multispecialty Research, Norfolk, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Premier Clinical Research, Spokane, Washington
- Australia (2):
  - Premier Specialists PTY LTD, Kogarah, New South Wales
  - Sinclair Dermatology, East Melbourne, Victoria
- Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubinsky MC, Wu J, McDonnell A, Lazin K, Goetsch M, Branquinho D, Modesto I, Armuzzi A. Low Incidence of Macular Edema and Other Ocular Events in the Etrasimod Development Program. J Crohns Colitis. 2025 May 8;19(5):jjae173. doi: 10.1093/ecco-jcc/jjae173. PMID 39575597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-treatment period study (12-Week Double-Blind Treatment Period and 52-Week Open-label extension [OLE] Period), to evaluate the safety and efficacy of etrasimod monotherapy compared with placebo in participants with moderate-to-severe atopic dermatitis (AD), whose disease was not adequately controlled with topical therapies.
Pre-assignment Details: A total of 140 participants were randomized into the 12-week Double-Blind Treatment Period and a total of 95 participants continued into the 52-Week OLE Period.
Groups:
- Double-blind Treatment Period: Etrasimod 1 Milligrams (mg): Participants with chronic AD were randomized to receive etrasimod 1 mg orally once daily for 12 weeks. Participants who successfully completed 12 weeks of Double-blind treatment continued to have access to etrasimod in the OLE period of the study.
- Double-blind Treatment Period: Etrasimod 2 mg: Participants with chronic AD were randomized to receive etrasimod 2 mg orally once daily for 12 weeks. Participants who successfully completed 12 weeks of Double-blind treatment continued to have access to etrasimod in the OLE period of the study.
- Double-blind Treatment Period: Placebo: Participants with chronic AD were randomized to receive placebo orally once daily for 12 weeks. Participants who successfully completed 12 weeks of Double-blind treatment continued to have access to etrasimod in the OLE period of the study.
- OLE Period: Etrasimod 2 mg: Participants who successfully completed 12 weeks of Double-blind treatment (who received etrasimod 1 mg, etrasimod 2 mg and placebo) continued to the OLE period and received etrasimod 2 mg orally once daily for 52 weeks. Participants who stopped taking study treatment before the end of the Double-blind Treatment period were not eligible to participate in the OLE Period.
Period: Double-blind Treatment (12-Week)
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo | OLE Period: Etrasimod 2 mg
Started | 47 | 47 | 46 | 0
Completed | 34 | 36 | 37 | 0
Not Completed | 13 | 11 | 9 | 0
Not completed — Adverse Event | 2 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 1 | 6 | 0
Not completed — Protocol deviation | 1 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0
Period: OLE Period (52-Week)
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo | OLE Period: Etrasimod 2 mg
Started | 0 | 0 | 0 | 95 (12 participants completed the Double-blind treatment period but did not enter the OLE Phase)
Completed | 0 | 0 | 0 | 68
Not Completed | 0 | 0 | 0 | 27
Not completed — Adverse Event | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 10
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 9
Not completed — Protocol deviation | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants, irrespective of whether they received any study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo | Total
Number analyzed (Participants) | 47 | 47 | 46 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (13.32) | 41.8 (14.83) | 44.1 (16.16) | 42.5 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 27 | 85
  Male | 17 | 19 | 19 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 26 | 31 | 84
  Asian | 2 | 3 | 2 | 7
  Black or African American | 15 | 18 | 11 | 44
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Treatment Period: Percent Change in Eczema Area and Severity Index (EASI) Score
Description: EASI evaluates severity of participant's AD based on severity of AD clinical signs and percent (%) of body surface area (BSA) affected. EASI is a composite scoring assessment of the affected area in 4 specific disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification), which was each assessed on a scale of "0" (absent) through "3" (severe). The EASI Area Score is documented for 4 regions of the body. Region 1: head and neck; Region 2: trunk (including genital area); Region 3: upper limbs; and Region 4: lower limbs (including buttocks), with the area of AD involvement assessed as a percentage by body area and converted to a score of 0 to 6. Total EASI score ranged from 0 to 72; higher score indicated greater severity of AD. Baseline is defined as Day 1 pre-randomization assessments.
Time Frame: Baseline (Day 1) and Week 12
Population: Full Analysis Set Population
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 47 | 47 | 46
Percent change | -58.68 (7.735) | -57.18 (7.800) | -48.41 (8.378)
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.1198, ANCOVA; Least square mean difference = -10.28, 95% CI 2-sided [-23.228 to 2.674], Standard Error of Mean 6.605
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Etrasimod 2 mg vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.1783, ANCOVA; Least square mean difference = -8.77, 95% CI 2-sided [-21.544 to 4.002], Standard Error of Mean 6.515

2. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants Achieving EASI-75
Description: EASI-75 is defined as a 75% reduction or greater in EASI score from Baseline to Week 12. Baseline is defined as Day 1 pre-randomization assessments.
Time Frame: Baseline (Day 1) and Week 12
Population: Full Analysis Set Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 47 | 47 | 46
Percentage of participants | 27.7 [15.62 to 42.64] | 38.3 [24.51 to 53.62] | 26.1 [14.27 to 41.13]
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.9826, Cochran-Mantel-Haenszel; Response Rate Difference = -0.2, 95% CI 2-sided [-18.52 to 18.11], Standard Error of Mean 9.34
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Etrasimod 2 mg vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.1891, Cochran-Mantel-Haenszel; Response Rate Difference = 13.0, 95% CI 2-sided [-6.12 to 32.21], Standard Error of Mean 9.78

3. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants Achieving a Validated Investigator Global Assessment (vIGA) 0 or 1 Score and a Reduction From Baseline of >= 2 Points
Description: The vIGA scale for AD is a 5-point scale to measure disease severity. The vIGA score was selected using descriptors that best described the overall appearance of skin lesions at a given time point using the following scoring: 0 = clear (no inflammatory signs of AD); 1 = almost clear (barely perceptible erythema and papulation); 2 = mild (slight but definite erythema and papulation); 3 = moderate (clearly perceptible erythema and papulation); and 4 = severe (marked erythema and papulation); Higher score indicated greater severity. Baseline is defined as Day 1 pre-randomization assessments.
Time Frame: Baseline (Day 1) and Week 12
Population: Full Analysis Set Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 47 | 47 | 46
Percentage of participants | 14.9 [6.20 to 28.31] | 29.8 [17.34 to 44.89] | 13.0 [4.94 to 26.26]
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.7694, Cochran-Mantel-Haenszel; Response Rate Difference = 2.2, 95% CI 2-sided [-12.29 to 16.64], Standard Error of Mean 7.38
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Etrasimod 2 mg vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.0450, Cochran-Mantel-Haenszel; Response Rate Difference = 17.4, 95% CI 2-sided [0.79 to 34.00], Standard Error of Mean 8.47

4. Secondary Outcome: Double-blind Treatment Period: Percent Change in Weekly Peak Pruritus Numerical Rating Scale (NRS) From an Itch Daily Diary
Description: Pruritus NRS is an assessment tool that was used to report the intensity of a participant's pruritus (itch). The scale for the pruritus NRS ranged from 0 to 10 with 0 being "no itch" and 10 being "the worst itch imaginable; higher scores indicated greater severity. Baseline is defined as Day 1 pre-randomization assessments.
Time Frame: Baseline (Day 1) and Week 12
Population: Full Analysis Set Population. Only those participants with data available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 27 | 32 | 31
Percent change | -38.401 (8.236) | -35.044 (7.910) | -24.374 (8.492)
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.0558, Mixed Models Analysis; Least square mean difference = -14.03, 95% CI 2-sided [-28.406 to 0.352], Standard Error of Mean 7.295
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Etrasimod 2 mg vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.1363, Mixed Models Analysis; Least square mean difference = -10.67, 95% CI 2-sided [-24.737 to 3.397], Standard Error of Mean 7.134

5. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants With Improvement (Reduction) in Peak Pruritus NRS Greater Than or Equal to (>=)3 From an Itch Daily Diary
Description: Pruritus NRS is an assessment tool that was used to report the intensity of a participant's pruritus (itch). The scale for the pruritus NRS ranged from 0 to 10 with 0 being "no itch" and 10 being "the worst itch imaginable; higher scores indicated greater severity. Percentage of participants with improvement (reduction) in peak pruritus NRS >=3 from an itch daily diary is presented. Baseline is defined as Day 1 pre-randomization assessments.
Time Frame: Baseline (Day 1) and Week 12
Population: Full Analysis Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 40 | 40 | 39
Percentage of participants | 45.0 [29.26 to 61.51] | 45.0 [29.26 to 61.51] | 41.0 [25.57 to 57.90]
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.7143, Cochran-Mantel-Haenszel; Response Rate Difference = 4.2, 95% CI 2-sided [-18.00 to 26.41], Standard Error of Mean 11.33
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Etrasimod 2 mg vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.6488, Cochran-Mantel-Haenszel; Response Rate Difference = 5.1, 95% CI 2-sided [-16.62 to 26.87], Standard Error of Mean 11.09

6. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants Achieving EASI-50
Description: EASI-50 is defined as a 50% reduction or greater of EASI from Baseline to Week 12. Percentage of participants achieving EASI-50 is presented. Baseline is defined as Day 1 pre-randomization assessments.
Time Frame: Baseline (Day 1) and Week 12
Population: Full Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 47 | 47 | 46
Percentage of participants | 61.7 [46.38 to 75.49] | 66.0 [50.69 to 79.14] | 52.2 [36.95 to 67.11]
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.3981, Cochran-Mantel-Haenszel; Response Rate Difference = 8.8, 95% CI 2-sided [-11.27 to 28.80], Standard Error of Mean 10.22
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Etrasimod 2 mg vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.1410, Cochran-Mantel-Haenszel; Response Rate Difference = 15.2, 95% CI 2-sided [-4.72 to 35.15], Standard Error of Mean 10.17

7. Secondary Outcome: Double-blind Treatment Period: Percentage of Participants Achieving EASI-90
Description: EASI-90 is defined as as a 90% reduction or greater of EASI from Baseline to Week 12. Percentage of participants achieving EASI-90 is presented Baseline is defined as Day 1 pre-randomization assessments.
Time Frame: Baseline (Day 1) and Week 12
Population: Full Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 47 | 47 | 46
Percentage of participants | 19.1 [9.15 to 33.26] | 14.9 [6.20 to 28.31] | 10.9 [3.62 to 23.57]
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.2690, Cochran-Mantel-Haenszel; Response Rate Difference = 8.4, 95% CI 2-sided [-6.61 to 23.38], Standard Error of Mean 7.65
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Etrasimod 2 mg vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.5428, Cochran-Mantel-Haenszel; Response Rate Difference = 4.3, 95% CI 2-sided [-9.56 to 18.25], Standard Error of Mean 7.09

8. Secondary Outcome: Double-blind Treatment Period: Percent Change in Percent Body Surface Area (BSA)
Description: BSA affected by AD were assessed for each section of the body. The possible highest score for each region was: head and neck (9%), anterior trunk (18%), back (18%), upper limbs (18%), lower limbs (36%), and genitals (1%) and were reported as a percentage of all major body sections combined; higher % BSA indicated greater severity. Baseline is defined as Day 1 pre-randomization assessments
Time Frame: Baseline (Day 1) and Week 12
Population: Full Analysis Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo
Number analyzed (Participants) | 36 | 39 | 39
Percent change | -34.725 (7.047) | -45.153 (6.860) | -31.913 (7.012)
Statistical Analysis 1: Comparison: Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.7163, Mixed Models Analysis; Least square mean difference = -2.81, 95% CI 2-sided [-18.089 to 12.466], Standard Error of Mean 7.721
Statistical Analysis 2: Comparison: Double-blind Treatment Period: Etrasimod 2 mg vs Double-blind Treatment Period: Placebo; Week 12; Test type: Superiority; p = 0.0840, Mixed Models Analysis; Least square mean difference = -13.24, 95% CI 2-sided [-28.284 to 1.805], Standard Error of Mean 7.602

9. Secondary Outcome: Open-label Extension (OLE) Period: Percent Change in EASI
Description: EASI evaluates severity of participant's AD based on severity of AD clinical signs and percent (%) of body surface area (BSA) affected. EASI is a composite scoring assessment of the affected area in 4 specific disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification), which was each assessed on a scale of "0" (absent) through "3" (severe). The EASI Area Score is documented for 4 regions of the body. Region 1: head and neck; Region 2: trunk (including genital area); Region 3: upper limbs; and Region 4: lower limbs (including buttocks), with the area of AD involvement assessed as a percentage by body area and converted to a score of 0 to 6. Total EASI score ranged from 0 to 72; higher score indicated greater severity of AD. Baseline is defined as the last measurement prior to the first etrasimod dose started at Week 16.
Time Frame: Baseline (Week 16) and Week 68
Population: Safety Set Population included all randomized participants who received at least 1 dose of study intervention. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- OLE Period: Etrasimod 2 mg: Participants who successfully completed 12 weeks of Double-blind treatment (who received etrasimod 1 mg, etrasimod 2 mg and placebo) and continued to the OLE period received etrasimod 2 mg orally once daily for 52 weeks. Participants who stopped taking study treatment before the end of the Double-blind Treatment period were not eligible to participate in the OLE Period.
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 68
Percent change | -45.39 (258.796)

10. Secondary Outcome: OLE Period: Number of Participants Achieving a EASI-75 Score
Description: EASI evaluates severity of participant's AD based on severity of AD clinical signs and percent (%) of body surface area (BSA) affected. EASI is a composite scoring assessment of the affected area in 4 specific disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification), which was each assessed on a scale of "0" (absent) through "3" (severe). The EASI Area Score is documented for 4 regions of the body. Region 1: head and neck; Region 2: trunk (including genital area); Region 3: upper limbs; and Region 4: lower limbs (including buttocks), with the area of AD involvement assessed as a percentage by body area and converted to a score of 0 to 6. Total EASI score ranged from 0 to 72; higher score indicated greater severity of AD. EASI-75 is defined as a >=75% reduction or greater of EASI from Baseline.
Time Frame: Baseline (Week 16) and Week 68
Population: Safety Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 68
Participants | 65

11. Secondary Outcome: OLE Period: Number of Participants Achieving a Validated Investigator Global Assessment (vIGA) 0 or 1 Score and a Reduction From Baseline of ≥ 2 Points
Description: The vIGA scale for AD is a 5-point scale to measure disease severity. The vIGA score was selected using descriptors that best described the overall appearance of skin lesions at a given time point using the following scoring: 0 = clear (no inflammatory signs of AD); 1 = almost clear (barely perceptible erythema and papulation); 2 = mild (slight but definite erythema and papulation); 3 = moderate (clearly perceptible erythema and papulation); and 4 = severe (marked erythema and papulation); Higher score indicated greater severity.
Time Frame: Baseline (Week 16) and Week 68
Population: Safety Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 69
Participants | 31

12. Secondary Outcome: OLE Period: Percent Change in SCORing Atopic Dermatitis (SCORAD) Total Score
Description: The SCORAD is a validated measure of the extent and severity of AD using 3 components: A = extent or affected BSA, B = severity and C = subjective symptoms. The extent of AD was assessed as percentage of each defined body area and reported as the sum of all areas, with a maximum score of 100%. The severity of 6 specific symptoms was assessed using the following scale: none (0), mild (1), moderate (2), or severe (3) (for a maximum of 18 total points, assigned as "B" in the overall SCORAD calculation). Subjective assessment of itch and sleeplessness was recorded for each symptom by the participant or relative on a Visual Analogue Scale, where 0 is no itch (or sleeplessness) and 10 is the worst imaginable itch (or sleeplessness), with a maximum possible score of 20. This parameter is assigned as "C" in the overall SCORAD calculation. The total SCORAD ranged from 0 (no disease) to 103 (severe disease); higher score indicated more severe AD.
Time Frame: Baseline (Week 16) and Week 68
Population: Safety Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 68
Percent change | -64.27 (69.273)

13. Secondary Outcome: OLE Period: Percent Change in Percent BSA
Description: BSA affected by AD were assessed for each section of the body. The possible highest score for each region was: head and neck (9%), anterior trunk (18%), back (18%), upper limbs (18%), lower limbs (36%), and genitals (1%) and were reported as a percentage of all major body sections combined; higher % BSA indicated greater severity. Baseline is defined as the last measurement prior to the first etrasimod dose started at Week 16.
Time Frame: Baseline (Week 16) and Week 68
Population: Safety Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 68
Percent change | -68.47 (52.083)

14. Secondary Outcome: OLE Period: Percent Change in Weekly Peak Pruritus NRS From an Itch Daily Diary
Description: Pruritus NRS is an assessment tool that was used to report the intensity of a participant's pruritus (itch). The scale for the pruritus NRS ranged from 0 to 10 with 0 being "no itch" and 10 being "the worst itch imaginable; higher scores indicated greater severity. Baseline is defined as the last measurement prior to the first etrasimod dose started at Week 16.
Time Frame: Baseline (Week 16) and Week 28
Population: Safety Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 56
Percent change | -36.87 (45.219)

15. Secondary Outcome: OLE Period: Change in Patient-Oriented Eczema Measure (POEM)
Description: The POEM is a participant-derived validated tool used for monitoring atopic eczema severity. The POEM consisted of 7 questions asking participants to rank how many days over the past 7 days they had experienced specific AD-related symptoms. Each of the 7 questions carried equal weight and was scored from 0 to 4 as follows: No days = 0; 1-2 days = 1; 3-4 days = 2; 5-6 days = 3; Every day = 4. The scores from the 7 questions were added up to give an overall POEM score as: 0-2 = 'clear/almost clear', 3-7 = 'mild', 8-16 = 'moderate', 17-24 = 'severe', and 25-28 = 'very severe atopic eczema'; higher scores indicated worse atopic eczema severity. Baseline is defined as the last measurement prior to the first etrasimod dose started at Week 16.
Time Frame: Baseline (Week 16) and Week 68
Population: Safety Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 65
Scores on a scale | -6.3 (6.50)

16. Secondary Outcome: OLE Period: Change in Dermatology Life Quality Index (DLQI)
Description: The DLQI is a validated 10-item questionnaire designed to measure the impact of skin disease on the Quality of Life (QoL). DLQI is a response to 10 items, which assessed QoL over the past week. For each item, the scale was rated as follows: 0 = "not at all"; 1 = "a little"; 2 = "a lot"; 3 = "very much," with an overall scoring system of 0 to 30; higher scores indicated a poor QoL. Baseline is defined as the last measurement prior to the first etrasimod dose started at Week 16.
Time Frame: Baseline (Week 16) and Week 68
Population: Safety Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 65
Scores on a scale | -5.4 (6.03)

17. Secondary Outcome: OLE Period: Change in Patient Global Assessment (PGA) of Disease
Description: PGA is an assessment tool that was used by participant to rate the disease and disease severity. Participants rated their overall well-being based on a 5-point Likert scale from poor to excellent. Response choices were: 1- 'Poor', 2- 'Fair', 3- 'Good', 4- 'Very Good,' or 5- 'Excellent'; higher scores indicated better well-being. For the 5-point Likert scale, a positive change from baseline indicates an improvement. Baseline is defined as the last measurement prior to the first etrasimod dose started at Week 16.
Time Frame: Baseline (Week 16) and Week 68
Population: Safety Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | OLE Period: Etrasimod 2 mg
Number analyzed (Participants) | 65
Scores on a scale | 1.23 (1.209)

ADVERSE EVENTS:
Time Frame: All-cause mortality, TEAEs and SAEs were collected for Double-blind Treatment period (12-Week) and for OLE Period (52-Week).
Description: Safety Population
Arm/Group | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) | Double-blind Treatment Period: Etrasimod 2 mg | Double-blind Treatment Period: Placebo | OLE Period: Etrasimod 2 mg
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/46 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/46 | 3/95
Other Adverse Events (participants affected / at risk) | 19/47 | 31/47 | 22/46 | 53/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) (N=47) | Double-blind Treatment Period: Etrasimod 2 mg (N=47) | Double-blind Treatment Period: Placebo (N=46) | OLE Period: Etrasimod 2 mg (N=95)
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Period: Etrasimod 1 Milligrams (mg) (N=47) | Double-blind Treatment Period: Etrasimod 2 mg (N=47) | Double-blind Treatment Period: Placebo (N=46) | OLE Period: Etrasimod 2 mg (N=95)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Eyelid cyst (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 4
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 2 | 0
Infection parasitic (Infections and infestations) | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 3 | 3
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ear canal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 1
Coagulation factor increased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Full blood count abnormal (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 2
Lymphocyte count decreased (Investigations) | 1 | 7 | 0 | 7
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 0 | 1
Red blood cells urine positive (Investigations) | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 5
Transaminases increased (Investigations) | 1 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 4
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 4 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 5
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT04162769/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04162769/SAP_001.pdf